CLINICAL TRIAL: NCT06329869
Title: A Phase II Study of Sacituzumab Govitecan for Advanced Esophageal Squamous Cell Carcinoma Patients
Brief Title: Sacituzumab Govitecan for Advanced Esophageal Squamous Cell Carcinoma
Acronym: SG-ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202401158MIFD
Record Dates: First submitted 2024-03-17; First posted 2024-03-26 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: sacituzumab govitecan; Trop-2
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab govitecan (Experimental)
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — Sacituzumab govitecan, 10 mg/kg intravenous infusion (the first infusion is to be administered over 3 hours; subsequent infusions may be administered over 1 to 2 hours if previous infusions were well tolerated) on day 1 and 8 of 21-day cycle.

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of sacituzumab govitecan in patients with advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Overexpression of Trop-2 was detected in ESCC compared with esophageal dysplasia. The investigators hypothesize that sacituzumab govitecan, by targeting Trop-2 which has been reported to be overexpressed in esophageal squamous cell carcinoma tumors, should have significant clinical activity in patients with advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients, 18 years of age or older, able to understand and give written informed consent.
2. Histologically proven squamous cell carcinoma of esophagus.
3. Patients with advanced ESCC, defined as those with unresectable locally advanced, recurrent, or metastatic disease, failed prior platinum-based chemotherapy and anti-PD-1/PD-L1 therapy (adjuvant anti-PD-1 therapy considered as prior exposure of anti-PD-1/PD-L1 therapy; progression or recurrence within 6 months of platinum-based chemoradiotherapy for localized disease considered as failed prior platinum-based chemotherapy).
4. Measurable disease as determined by RECIST 1.1. Lesions in previously irradiated areas should not be considered measurable unless they have progressed since the radiotherapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
6. Archival tumor tissue for Trop-2 expression and optional fresh biopsy if feasible.
7. Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation (hemoglobin ≥ 9 g/dL, ANC ≥ 1500/mm3, and platelets ≥ 100,000/µL).
8. Adequate hepatic function (bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN if known liver metastases, and serum albumin > 3 g/dL).
9. Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation {Cockcroft 1976}.
10. Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception as described in Appendices.
11. Willing and able to comply with the requirements and restrictions in this protocol.

Exclusion Criteria:

1. Positive serum pregnancy test or women who are breastfeeding.
2. Known hypersensitivity to the study drug, its metabolites, or formulation excipient.
3. Requirement for ongoing therapy with or prior use of any prohibited medications.
4. Have had a prior anticancer biologic agent within 4 weeks prior to enrollment or have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to enrollment and have not recovered (ie, ≥ Grade 2 is considered not recovered) from AEs at the time of study entry.
5. Have not recovered (ie, ≥ Grade 2 is considered not recovered) from AEs due to a previously administered agent. Patients with any grade neuropathy or alopecia are an exception to this criterion and will qualify for the study. If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Have previously received topoisomerase 1 inhibitors.
7. Have an active second malignancy. Patients with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumors with low risk of recurrence (eg, nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed.
8. Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment.
9. Have active serious infection requiring antibiotics.
10. Have known history of HIV-1 or 2 (or positive HIV-1/2 antibody, if done at screening) with detectable viral load or taking medications that may interfere with SN-38 metabolism.
11. Have active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.

    1. Patients who test positive for hepatitis B surface antigen (HBsAg) will not be eligible. Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
    2. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease.
12. Patients who test positive for HIV antibody.
13. Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
14. Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the patient's participation in the study.
15. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of study drug.
16. No adequate archival or fresh ESCC tumor tissues for characterization of Trop-2 expression.
17. Active central nervous system metastases.
18. Adenocarcinoma of esophagus or gastroesophageal junction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Overall objective response rates (ORR) | 18 weeks
  The proportion of patients whose tumor response is categorized as complete response (CR) and partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
  The time from enrollment to death of any cause or the last follow-up (censored).
Progression-free survival (PFS) | 6 months
  The time from enrollment to the first occurrence of disease progression or death from any cause (whichever occurs first) and will be conducted in the whole study population.
Duration of response (DOR) | 6 months
  The time measurement criteria are ﬁrst met for CR/PR (whichever is ﬁrst recorded) until the ﬁrst date that progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 months
  Toxicities per CTCAE 5.0

OTHER OUTCOMES:
Biomarkers-related endpoints | 18 weeks
  ORR by RECIST 1.1 according to immunohistochemistry-(IHC)-detected Trop-2 expression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No